CLINICAL TRIAL: NCT03592654
Title: Pilot Study: A Telehealth Intervention for Caregivers of Infants With Early Signs of Autism Spectrum Disorder- Infant TeleHelp Study
Brief Title: Pilot Study: A Telehealth Intervention for Caregivers of Infants With Early Signs of Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1249018
Record Dates: First submitted 2018-06-25; First posted 2018-07-19 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Autism Spectrum Disorder; Developmental Delay
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Intervention Model Description: single subject multiple baseline design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- infant telehelp condition (Experimental): caregiver coaching to improve infant behaviors that indicate they are at risk for autism spectrum disorder
  Interventions: Behavioral: infant telehelp

INTERVENTIONS:
Behavioral: infant telehelp — Adapted from Early Start Denver Model (ESDM), a naturalistic developmental behavioral intervention

SUMMARY:
Caregiver coaching will be provided using telehealth technology, in order to determine the efficacy and effectiveness of the telehealth medium of intervention delivery for caregivers of infants with concern for ASD.

DETAILED DESCRIPTION:
Ideally, all caregivers with an infant identified with concern for ASD would have immediate access to good quality caregiver coaching provided in the most natural environment possible. However, this is currently not the case for the majority of families. There are no empirically validated treatment programs for infants showing ASD risk. The proposed research project will use Applied Behavior Analysis-based single-subject experimental designs to further develop a promising caregiver-mediated intervention designed for infants showing early signs of ASD. Caregiver coaching will be provided using telehealth technology, in order to maximize recruitment opportunities and to determine the efficacy and effectiveness of the telehealth medium of intervention delivery for caregivers of infants with concern for ASD.

ELIGIBILITY:
Inclusion Criteria:

* Infants must exhibit early symptoms of ASD as indicated by a combination of Autism Observation Scale for Infants (AOSI) scores of 7 or higher
* and Infant Toddler Checklist (ITC) scores in the autism concern range
* Expression of clinical concern about ASD risk by the assessor and caregiver
* Caregivers must be identified as the infants' primary caregivers
* Caregivers be English speaking
* Caregivers must have access to wired or wireless network technology to access the internet in their homes.

Exclusion Criteria:

* Infants may not have had significant abnormalities in the pre-, peri-, and postnatal period or gestational age younger than 34 weeks
* Infants may not have serious medical conditions involving repeated or lengthy hospitalizations, head injuries, seizures, cerebral palsy or impaired hand use
* Infants may not have multiple daily administrations of medical treatment (e.g., nebulizers daily)
* Infants may not have known genetic syndrome associated with ASD (e.g., fragile X syndrome) Infants may not have moderate to severe visual, auditory, or motor impairments
* A caregiver may be excluded from participation if the caregiver is engaging in the majority of all possible caregiver treatment target behaviors at therapeutic levels during intake (Fidelity of Implementation scores of 80% or higher on each caregiver target behavior).

Ages: 5 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Child Behaviors Targeted by Intervention | 7 months
  Treatment-targeted child behaviors (e.g., visual fixations on objects, abnormal repetitive behaviors, lack of age-appropriate phonemic development, lack of coordination of gaze, affect, and voice in reciprocal, turn-taking interactions) will be coded from 10-minute caregiver-infant dyad intervention video probes taken throughout all phases of the study.

SECONDARY OUTCOMES:
Autism Observation Scale for Infants | 7 months
  (AOSI; Bryson et al., 2006) The AOSI will be administered by caregivers at intake and exit. During the AOSI, infants are engaged in semi-structured play and systematic presses are designed to assess various target behaviors, including visual tracking and attention disengagement, coordination of eye gaze and action, imitation, affective responses, early social-communicative behaviors, behavioral reactivity, and sensory-motor development.
Ages and Stages Questionnaires, 3rd Edition | 7 months
  (ASQ-3; Squires & Bricker, 2015) The ASQ-3 are a series of questionnaires completed by a child's caregiver designed to assess the developmental performance of infants and children ages 1-66 months across five developmental areas: communication, gross motor, fine motor, problem solving, and personal-social. The ASQ-3 takes approximately 15 minutes to be completed.
Individual Growth and Development Indices | 7 months
  (IGDIs; Carta et al., 2010) IGDIs were developed to gather very frequent assessment of child developmental progress. We will use the Early Communication Index, ECI, and the Early Problem Solving Index, EPSI, domains appropriate for ages 5 to 50 mos. Two 6-minute semi-structured and video recorded play procedures will be carried out at intake and exit.
Vineland Adaptive Behavior Scales, 2nd edition | 7 months
  (VABS-II; Sparrow et al., 2005) The VABS-II consists of four domains of adaptive behavior: communication, self-care, social, and motor skills. The VABS-II is a semi-standardized caregiver questionnaire or interview designed to assess children's behavior in real life, everyday settings.
Parent Satisfaction Rating | 7 months
  (Charlop-Christy & Carpenter, 2000) This is a measure of social validity, or acceptability, of the experimental treatment, to caregivers. This scale will be administered to the caregivers at intake and exit. This tool allows caregivers to rate the ease of implementation in the home and their opinions concerning treatment utility.
Working Alliance Scale for Interventions with Children | 7 months
  (Davis et al., 2006). These measures will be administered to the caregivers at intake and exit and will be used to describe the response of the families to the experimental intervention, and thus constitutes another measure of social validity.
Caregiver Fidelity of Treatment Implementation | 7 months
  Caregiver fidelity of implementation (FI) of the Infant Start intervention will be coded from 10-minute caregiver-child dyad intervention video probes to determine caregivers' FI of intervention techniques over the course of the study. The fidelity tool involves having experts in Infant Start rate caregiver use of each of the intervention strategies on a 1-5 Likert rating scale, with a code of "1" meaning the caregiver did not implement the technique throughout the session and a code of "5" meaning the caregiver implemented the technique correctly throughout the session.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Dufek, PhD, Principal Investigator — UC Davis
Locations (1):
- MIND institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No